CLINICAL TRIAL: NCT02874248
Title: A Randomized, Double-blind, Placebo-controlled, Parallel, Single Center Study to Investigate the Pharmacokinetics, Safety, Tolerability, and QT Concentration-effect Modelling of Estetrol in Combination With Drospirenone After Single and Multiple Dosing in Healthy Women
Brief Title: E4/DRSP Single and Multiple Dose PK and Early QT Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MIT-Es0001-C103; 2016-000861-22 (EudraCT Number)
Record Dates: First submitted 2016-08-09; First posted 2016-08-22 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2016-08

CONDITIONS: Contraception
MeSH Terms: interventions — Estetrol; drospirenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group 1: 15 mg E4/3 mg DRSP (n=10) (Active Comparator): a single oral dose of 15 mg E4/3 mg DRSP (n=10) followed, after a washout of at least 14 days, by multiple oral doses of 15 mg E4/3 mg DRSP (n=10) once daily for 14 days
  Interventions: Drug: 15 mg E4/3 mg DRSP
- Group1: Placebo (n=4) (Placebo Comparator): a single oral dose of a placebo which visually matches the active medication, followed, after a washout of at least 14 days, by multiple oral doses of matching placebo once daily for 14 days
  Interventions: Drug: Visually matching placebo
- Group 2: 30 mg E4/6 mg DRSP (n=10) (Active Comparator): a single oral dose of 30 mg E4/6 mg DRSP, followed, after a washout of at least 14 days, by multiple oral doses of 30 mg E4/6 mg DRSP once daily for 14 days
  Interventions: Drug: 30 mg E4/6 mg DRSP
- Group 2: Placebo (n=4) (Experimental): a single oral dose of a placebo which visually matches the active medication, followed, after a washout of at least 14 days, by multiple oral doses of matching placebo once daily for 14 days
  Interventions: Drug: Visually matching placebo
- Group 3: 60 mg E4/12 mg DRSP (n=10) (Active Comparator): a single oral dose of 60 mg E4/12 mg DRSP, followed, after a washout of at least 14 days, by oral doses of 60 mg E4/12 mg DRSP once daily for 14 days
  Interventions: Drug: 60 mg E4/12 mg DRSP
- Group 3: Placebo (n=4) (Placebo Comparator): a single oral dose of a placebo which visually matches the active medication, followed, after a washout of at least 14 days, by multiple oral doses of matching placebo once daily for 14 days
  Interventions: Drug: Visually matching placebo
- Group 4: 75 mg E4/15 mg DRSP (n=9) (Active Comparator): a single oral dose of 75 mg E4/15 mg DRSP, followed, after a washout of at least 14 days, by oral doses of 75 mg E4/15 mg DRSP once daily for 14 days
  Interventions: Drug: 75 mg E4/15 mg DRSP
- Group 4: Placebo (n=4) (Placebo Comparator): a single oral dose of a placebo which visually matches the active medication, followed, after a washout of at least 14 days, by multiple oral doses of matching placebo once daily for 14 days
  Interventions: Drug: Visually matching placebo

INTERVENTIONS:
Drug: 15 mg E4/3 mg DRSP — a single oral dose of 15 mg E4/3 mg DRSP (n=10) followed, after a washout of at least 14 days, by multiple oral doses of 15 mg E4/3 mg DRSP (n=10) once daily for 14 days
  Other Names: 15 mg estetrol and 3 mg drospirenone
  Arms: Group 1: 15 mg E4/3 mg DRSP (n=10)
Drug: 30 mg E4/6 mg DRSP — a single oral dose of 30 mg E4/6 mg DRSP, followed, after a washout of at least 14 days, by multiple oral doses of 30 mg E4/6 mg DRSP once daily for 14 days
  Other Names: 30 mg estetrol and 6 mg drospirenone
  Arms: Group 2: 30 mg E4/6 mg DRSP (n=10)
Drug: 60 mg E4/12 mg DRSP — a single oral dose of 60 mg E4/12 mg DRSP, followed, after a washout of at least 14 days, by oral doses of 60 mg E4/12 mg DRSP once daily for 14 days
  Other Names: 60 mg estetrol and 12 mg drospirenone
  Arms: Group 3: 60 mg E4/12 mg DRSP (n=10)
Drug: Visually matching placebo — a single oral dose of a placebo which visually matches the active medication, followed, after a washout of at least 14 days, by multiple oral doses of matching placebo once daily for 14 days
  Arms: Group 2: Placebo (n=4); Group 3: Placebo (n=4); Group 4: Placebo (n=4); Group1: Placebo (n=4)
Drug: 75 mg E4/15 mg DRSP — a single oral dose of 75 mg E4/15 mg DRSP, followed, after a washout of at least 14 days, by oral doses of 75 mg E4/15 mg DRSP once daily for 14 days
  Arms: Group 4: 75 mg E4/15 mg DRSP (n=9)

SUMMARY:
This study is conducted to evaluate the effect of single and multiple therapeutic and supratherapeutic oral doses of E4/DRSP combinations on PK parameters, safety, tolerability and on cardiac repolarization, as detected by QT interval corrected with Fridericia's formula (QTcF).

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel, single center study in healthy female subjects. A total of 42 female subjects will be enrolled in 3 groups of 14 subjects each. A potential fourth group of 14 healthy female subjects may be added. In each group, subjects will be randomized in a 2.5 to 1 ratio between active (n=10) and placebo (n=4).

Subjects will receive a single dose on Day 1 and, after a washout of at least 14 days, multiple doses on 14 consecutive days from Days 15 to 28.

Group 1 and Group 2 may be dosed in parallel. After completion of Group 1 and Group 2, a Dose Escalation Report (DER), including PK data up to at least 24 hours post-last dose, will be prepared by the Principal Investigator (PI). Escalation to the planned dose level of 60 mg E4/12 mg DRSP will only proceed if the safety and tolerability of the dose levels of 15 mg E4/3 mg DRSP and 30 mg E4/6 mg DRSP up to 24 hours post-last dose, are acceptable to the PI and the Sponsor and, if deemed necessary by the Independent Ethics Committee (IEC) following their review of the protocol, after a statement of no objection of the DER from the IEC.

After completion of Group 3, a second DER, including PK data, will be prepared by the PI. If in Group 3 the expected exposure level of approximately 4 times the exposure of Group 1 is not achieved, and treatment in Group 3 is well tolerated, an additional group with 14 subjects may be enrolled, using a dose level that is estimated to result in at least 4 times the exposure after administration of the 15 mg E4/3 mg DRSP therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

1. Gender : Healthy female subject
2. Age : 18-50 years, inclusive
3. Body mass index (BMI) : 18.0-35.0 kg/m2
4. At screening, female subjects must be non-pregnant and non-lactating, or of non-childbearing potential
5. Willing to use a double-barrier method of contraception from screening until 90 days after the follow up visit.
6. Willingness to abstain from alcohol and grapefruit (juice) from 48 hours prior to admission into the clinical research center up to follow-up.
7. Normal resting supine blood pressure and pulse showing no clinically relevant deviations as judged by the PI at screening.
8. Computerized (12-lead) ECG recording without signs of clinically relevant pathology at screening
9. Willing and able to sign the ICF.
10. Willing and able to comply with the study procedures

Exclusion Criteria:

1. Postmenopausal status
2. History or presence of clinically relevant disease of any major system organ class (e.g., cardiovascular, pulmonary, renal, hepatic, gastrointestinal, reproductive, endocrinological, neurological, psychiatric or orthopedic disease) as judged by the PI
3. Condition of hyperkalemia resulting from renal insufficiency, hepatic dysfunction, adrenal insufficiency or medication intake
4. Previous participation in the current study
5. Use of:

   * combined contraceptives (i.e., COC, Nuvaring®) within 28 days prior to the first dose administration until study completion
   * progestogen-only contraceptive methods (e.g., minipill, implant, or hormonal intrauterine system) within 28 days prior to the first dose administration until study completion
   * depot progestogen preparations or an injectable hormonal method of contraception (e.g., Depo-Provera®) within 6 months prior to the first dose until study completion
6. Use of:

   * any prescription drugs or herbal supplements acting on CYP3A4 functions (e.g., St. John's Wort) within 28 days prior to the first study dose administration until study completion
   * any over-the-counter medication or dietary supplements (vitamins included) within 14 days prior to the first study dose administration until study completion.
7. Use of any tobacco products within the last 3 months prior to the first admission
8. History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
9. Positive drug screening
10. Positive screen for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) 1 and 2 antibodies
11. Participation in an investigational drug study within 60 days prior to the first drug administration in the current study
12. History of relevant drug and/or food allergies
13. Donation or loss of more than 100 mL of blood within 60 days prior to the first drug administration. Donation or loss of more than 1.0 L of blood in the 10 months prior to the first drug administration in the current study
14. Significant and/or acute illness within 5 days prior to the first drug administration that may impact safety assessments, as judged by the PI
15. History and/or family history of congenital long QT syndrome, unexplained syncope or other additional risks for Torsade de Pointes, or sudden death
16. History or presence of hormone-related malignancy treated or not, whatever the time of onset. History of malignancy of any other organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years prior to screening
17. History of migraine with aura
18. Any surgical or medical condition that could significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study
19. Contraindications for the use of contraceptive steroids
20. Sponsor employees or clinical site personnel directly affiliated with this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum observed plasma concentration of E4 and DSRP | On day 1 and day 28 (steady state)
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
Tmax: time to attain maximum observed plasma concentration of E4 and DSRP | On day 1 and day 28 (steady state)
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
AUC0-t: Area under the plasma concentration-time curve up to time t, where t is the last point with concentrations above the lower limit of quantitation (LLOQ) - for E4 and DSRP | On day 1 and day 28 (steady state)
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
AUC0-24: area under the plasma concentration-time curve up to time 24 hours (where 24 hours is the dosing interval) using linear-log trapezoidal rule - for E4 and DSRP | On day 1 only
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
AUC0-inf: Area under the plasma concentration-time curve from time 0 to infinity calculated as: AUC0-inf = AUC0-t + Clast/kel, where Clast is the last measurable plasma concentration | On day 1 only
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
Kel: terminal elimination rate constant of E4 and DSRP | On day 1 and day 28 (steady state)
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
T1/2: terminal elimination half-life of E4 and DSRP, calculated as 0.693/kel | On day 1 and day 28 (steady state)
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
AUC0-tau: Area under the plasma concentration time curve over a dosing interval tau - of E4 and DSRP | On day 28 only
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35
Ra: Accumulation ratio for AUC | On day 1 and day 28 (steady state)
  PK sampling on day 1, 2-3, 4-8, 16-25, 26-27, 28, 29, 30, 31-35

SECONDARY OUTCOMES:
Number of adverse events and number of subjects with AEs as a measure of safety and tolerability | From admission until follow-up visit (between day 37 and 41)
  Any clinically significant observations in results of clinical laboratory tests, 12-lead ECGs, echocardiography, continuous cardiac monitoring (Holter monitoring), vital signs, or physical examinations will be recorded as AEs
deltaQTcF as measured by Holter monitoring (continuous cardiac monitoring) | Time matched on day -1 (for baseline measurements) and on day 28: 1 hour pre-dose until 24h post-dose
  To define the effect of E4 in combination with DRSP on QT interval corrected with Fridericia's formula (QTcF)
ECG parameters | Once during screening period; on day -2, 2, 15, 28, 29; once between day 2-3 and once between day 37 and 41 (follow-up)
  To define the effect of E4 in combination with DRSP on heart rate (HR), PR, and QRS

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van de Wetering, MD, Principal Investigator — PRA Health Sciences

IPD SHARING:
Plan to Share IPD: No